CLINICAL TRIAL: NCT07186361
Title: Remote Symptom Assessment And Management Via Mobile App For Adults With Chronic Kidney Disease Living In Vietnam
Brief Title: Symptom Assessment And Management For Adults With CKD In Vietnam
Acronym: SAM-CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Griffith University (Other)
Responsible Party: Principal Investigator, Khanh Linh Bui, PhD Candidate, Griffith University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 135/2025/CN/HDDD VMEC
Record Dates: First submitted 2025-09-01; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; CKD; Symptom management; mobile app; eHealth; randomised feasibility trial; Vietnam
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Symptom Assessment

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to either the intervention or control groups with allocation rate is 2:1 (2 in intervention group: 1 in control group)
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study intervention, neither the patients nor the researchers can be blinded. However, the Outcome Assessor who collects study outcome data will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (SAM-CKD group) (Experimental): The intervention group will be invited to use the SAM-CKD program for 6 weeks
  Interventions: Device: Symptom Assessment and Management Program (SAM-CKD) which is delivered via Smart Kidney mobile app
- Control group (No Intervention): Participants in the control group will receive usual care and they will be offered to use the intervention after the study completes

INTERVENTIONS:
Device: Symptom Assessment and Management Program (SAM-CKD) which is delivered via Smart Kidney mobile app — An intervention program delivered through a mobile app to support symptom assessment and management for adults with CKD. The SAM-CKD program has three components - introduction, symptom tracker and symptom management. A list of 17 common symptoms will be assessed. Users can self-assess symptoms and rate these according to the severity level (overwhelmingly, severely, moderately, slightly, and not at all). The SAM-CKD program will provide symptom management strategies based on symptoms reported by patients. The intervention's duration is 6 weeks.
  Arms: Intervention group (SAM-CKD group)

SUMMARY:
Adults with chronic kidney disease (CKD) have many symptoms that lower their quality of life and put a huge burden on the healthcare system. Recently, eHealth solutions have been introduced in chronic kidney disease care, helping with symptom management and improving patient outcomes. While symptom management via electronic health (eHealth) is emerging in other countries, it has not commenced in Vietnam. This study aims to develop and evaluate a remote symptom assessment and management program delivered through a mobile application for adults with CKD living in Vietnam to help them manage their symptoms. This is the first intervention program focusing on symptom assessment and management in Vietnam. By assessing and managing symptoms, adults with CKD can better self-manage their symptoms.

DETAILED DESCRIPTION:
Adults with CKD experience a wide range of symptoms that significantly impact their health-related quality of life and place a huge burden on the healthcare system. Mobile health app-based interventions for symptom assessment and management have the potential to alleviate the burden of CKD and improve patient outcomes. This study aims to develop and test a Symptom Assessment and Management (SAM-CKD) program embedded into a mobile app for adults with CKD living in Vietnam. A feasibility randomised trial will be designed in designed following the Consolidated Standards of Reporting Trials (CONSORT) statement extension for randomised pilot and feasibility trials to evaluate the feasibility, usability, acceptability, and potential effectiveness of symptoms and health-related quality of life. Adults with CKD grade 4 or 5 (including those on dialysis) will be randomly assigned to either the intervention or control groups. Informed by the Theory of Symptom Management, the intervention includes three main components: a general introduction to CKD symptoms, a symptom tracker, and symptom management strategies. The intervention group will use the program for 6 weeks to self-manage their symptoms. Primary outcomes are feasibility and acceptability, measured by eligibility rate, recruitment rate, retention and attrition, protocol adherence, mobile app usability and acceptability. Secondary outcomes are changes in CKD symptoms and health-related quality of life measured by Integrated Palliative Outcome Scale - Renal (IPOS-Renal) and European Quality of Life 5-Dimension 5-Level Questionnaire (EQ-5D-5L), respectively. Data analysis involves descriptive and intention-to-treat analyses. The results will be reported following the CONSORT statement extension for randomised pilot and feasibility trials. Findings will provide empirical evidence about the feasibility, acceptability and initial effectiveness of mobile-based symptom management intervention and will inform the design of future large-scale effectiveness studies.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* are diagnosed with CKD grade 4 or grade 5 with or without haemodialysis
* speak and read Vietnames
* own a smartphone operating on Android with internet accessibility
* agree to participate in this study.

Exclusion Criteria:

* cognitive impairment
* psychological problems
* terminal illness, such as cancer and advanced lung disease
* acutely unwell
* participating in another study during this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the SAM program (Eligibility) | Baseline (week 0)
  The eligibility rate will be calculated by dividing the number of eligible participants by the number of screened participants. The eligibility rate will be reported in percentage.
Usability and Acceptability | Week 6
  The usability and acceptability will be assessed after participants complete 6 weeks of intervention using the Vietnamese version of the Mobile App Usability Questionnaire. This is an 18-item self-rated measure of the usability and acceptability of mobile apps. It has three subscales: 1) ease of use (5 items), 2) interface and satisfaction (7 items), and 3) usefulness (6 items). Each item is rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The app's usability is determined by the total and average of all statements. The total score ranges from 18 to 126; the higher the overall total and average, the better the app's usability.
Feasibility of the SAM program (recruitment rate) | Baseline (week 0)
  The recruitment rate will be calculated by dividing the number of recruited participants by the number of eligible participants and reported as percentage.
Feasibility of the SAM program (attrition rate) | Week 6
  The attrition rate will be determined by the number of participants who drop out before completing the study and reported as percentage.
Feasibility of the SAM program (retention rate) | Week 6
  The retention rate will be calculated by the number of participants who complete the study by dividing the number of participants who enrolled. The retention rate will be reported in percentage.
Feasibility of the SAM program (protocol adherence) | Week 6
  The protocol adherence is the number of participants in the allocated group who receive the assigned intervention. The protocol adherence will be reported in percentage
Feasibility of the SAM program (missing data) | 3 time points (week 0, week 3, week 6)
  Missing data is the percentage of data missing from the study's reporting.

SECONDARY OUTCOMES:
Symptoms | 3 time points (week 0, week 3, and week 6)
  The Vietnamese version of Integrated Palliative Care Outcome Scale - Renal (IPOS-Renal) will be used to assess symptoms of participants in both groups. It has 11 items covering five components: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The last four items are about information needs, satisfaction with healthcare and practical issues. Items scored on a Likert scale from 0 to 4 for increasing severity; total score reflects symptom burden. The higher total score, the higher symptom burden.
Health-related quality of life | 3 time points (week 0, week 3, and week 6)
  Health-related quality of life will be assessed using a self-reported EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) Vietnamese version. The tool includes five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The lower score of each dimensions, the better patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Bonner, PhD, Principal Investigator — School of Nursing and Midwifery, Griffith University
Locations (1):
- E Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
All Individual participant data (IPD) that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months after publication with no end date
Access Criteria: The IPD can be assessed underlie a publication
URL: https://www.griffith.edu.au/

REFERENCES:
- [Background] Okpechi IG, Muneer S, Ye F, Zaidi D, Ghimire A, Tinwala MM, Saad S, Osman MA, Lunyera J, Tonelli M, Caskey F, George C, Kengne AP, Malik C, Damster S, Levin A, Johnson D, Jha V, Bello AK. Global eHealth capacity: secondary analysis of WHO data on eHealth and implications for kidney care delivery in low-resource settings. BMJ Open. 2022 Mar 23;12(3):e055658. doi: 10.1136/bmjopen-2021-055658. PMID 35321893
- [Background] Marin AE, Redolat R, Gil-Gomez JA, Mesa-Gresa P. Addressing Cognitive Function and Psychological Well-Being in Chronic Kidney Disease: A Systematic Review on the Use of Technology-Based Interventions. Int J Environ Res Public Health. 2023 Feb 14;20(4):3342. doi: 10.3390/ijerph20043342. PMID 36834042
- [Background] Zhang JC, El-Majzoub S, Li M, Ahmed T, Wu J, Lipman ML, Moussaoui G, Looper KJ, Novak M, Rej S, Mucsi I. Could symptom burden predict subsequent healthcare use in patients with end stage kidney disease on hemodialysis care? A prospective, preliminary study. Ren Fail. 2020 Nov;42(1):294-301. doi: 10.1080/0886022X.2020.1744449. PMID 32506997
- [Background] van Oevelen M, Bonenkamp AA, van Eck van der Sluijs A, Bos WJW, Douma CE, van Buren M, Meuleman Y, Dekker FW, van Jaarsveld BC, Abrahams AC; DOMESTICO study group. Health-related quality of life and symptom burden in patients on haemodialysis. Nephrol Dial Transplant. 2024 Feb 28;39(3):436-444. doi: 10.1093/ndt/gfad179. PMID 37580140
- [Background] Speyer E, Tu C, Zee J, Sesso R, Lopes AA, Moutard E, Omorou AY, Stengel B, Finkelstein FO, Pecoits-Filho R, de Pinho NA, Pisoni RL; CKDopps Investigators. Symptom Burden and Its Impact on Quality of Life in Patients With Moderate to Severe CKD: The International Chronic Kidney Disease Outcomes and Practice Patterns Study (CKDopps). Am J Kidney Dis. 2024 Dec;84(6):696-707.e1. doi: 10.1053/j.ajkd.2024.06.011. Epub 2024 Aug 6. PMID 39117097
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Derived] Bui KL, Hyun A, Purtell L, Hoang VL, Bonner A. Remote symptom assessment and management via mobile app for adults with chronic kidney disease in Vietnam (SAM-CKD programme): a randomised feasibility trial protocol. BMJ Open. 2026 Feb 6;16(2):e111934. doi: 10.1136/bmjopen-2025-111934. PMID 41651513

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT07186361/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT07186361/ICF_001.pdf